CLINICAL TRIAL: NCT00992108
Title: Efficacy of Botulinum Toxin Versus Lidocaine in Treating Masticatory Myofascial Face Pain Using Ultrasound and EMG Guided Techniques
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of eligible patients willing and able to participate
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8295968
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Results first posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-11

CONDITIONS: Face Pain
Keywords: Bruxism; Myofascial pain; EMG; Ultrasound; Masticatory myofascial face pain from bruxism and clenching
MeSH Terms: conditions — Facial Pain; Bruxism | interventions — Lidocaine; Nerve Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine (Active Comparator): lidocaine injection group
  Interventions: Drug: lidocaine
- Botulinum (Experimental)
  Interventions: Drug: chemodenervation

INTERVENTIONS:
Drug: lidocaine — 1cc 1%
  Arms: Lidocaine
Drug: chemodenervation — botulinum toxin
  Arms: Botulinum

SUMMARY:
Botulinum toxin-A (BTX-A) prevents the release of acetylcholine in presynaptic terminals of the neuromuscular junction. It has been proposed to be effective in spastic conditions of the head and neck including oromandibular dystonias, bruxism, and muscular hypertrophy (1,2,3,4). However, only one randomized, double-blinded, placebo controlled trial has been completed involving 20 patients demonstrating both objective and subjective improvement in the BTX-A treated group over those treated with saline at one week, one month, and six months (5).

Currently, in most orofacial pain practices, when the diagnosis of masticatory myofascial pain in the head region is made, patients are treated with a standard myofascial protocol. This protocol involves stretching, application of moist heat, spray and stretch, and lidocaine trigger point injections into the masticatory muscles. This is considered the standard of care among most orofacial pain practioners.

There have been no randomized, double-blinded, head-to-head trials comparing BTX-A injections to lidocaine injections in the treatment of masticatory myofacial pain. Moreover, in all studies, muscles were targeted using surface landmarks with no confirmatory tests to guarantee the medication was administered to the intended muscle. In previous studies, the medial and lateral pterygoid muscles, important masticatory muscles that is often hyperactive in masticatory myofacial pain was not injected due to lack of palpable surface landmarks. Ultrasound and electromyography (EMG) guidance will help us locate these muscles.

The purpose of this study is to objectively measure functional improvement in patients with masticatory myofascial pain injected with lidocaine versus BTX-A. A pilot study enrolling 20 patients is proposed. 20 patients will be randomized to receive either BTX-A or lidocaine injections into the bilateral temporalis, masseter, and medial and lateral pterygoid. Objective and subjective clinical parameters will be measured. These include pain at rest and with chewing, maximum non-assisted and assisted mouth opening, protrusive and laterotrusive jaw movements, subjective efficacy of treatment, and side-effects of treatment. Patients will be assessed at baseline, one week, one month, and three months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are to have identifiable painful myofascial trigger points in the masseter, temporalis, and medial and lateral pterygoid muscles.
* Subjects will be examined by the principle investigators to determine if the individual is a suitable candidate for the study, based on active trigger points and willingness to participate in the study

Exclusion Criteria:

* Pregnant woman will be excluded from participation as potential risk is noted in product label indications. Individuals over the age of 65 will be excluded per product label indications that reflect lack of data in individuals over age 65.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Chang, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- Westwood Associates, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lidocaine | Botulinum
Started | 7 | 10
Completed | 7 | 9
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine | Botulinum | Total
Number analyzed (Participants) | 7 | 10 | 17
Age, Continuous [Mean (Full Range); unit: years] | 57.14 [38 to 76] | 44.7 [24 to 65] | 49.82 [24 to 76]
Gender [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response as Assessed by >20% Change From Baseline in the Jaw Functional Limitation Scale (JFLS) Global Score
Description: The JFLS contains 20 items that measure limitations across mastication, vertical jaw mobility, and verbal/emotional expression rated on a 0-10 scale where 0 = "no limitation" and 10 = "severe limitation."
Time Frame: 4 months
Population: participants who completed the 4-month follow-up
Measure: Number; unit: participants
Arm/Group | Lidocaine | Botulinum
Number analyzed (Participants) | 7 | 9
participants | 5 | 7

2. Secondary Outcome: Clinical Response as Assessed by >20% Change From Baseline in the Jaw Functional Limitation Scale (JFLS) Global Score
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Lidocaine | Botulinum
Number analyzed (Participants) | 7 | 10
participants | 5 | 6

3. Secondary Outcome: Clinical Response as Assessed by >20% Change From Baseline in the Pressure Pain Threshold
Description: measurements were obtained by placing examiner's index finger of the examiner on the area of the trigger point (hyperirritable areas on skeletal muscle with palpable taut bands of muscle fibers) and exerting pressure until there was whitening of the nail bed. Pressure pain levels were rated subjectively by the participant and coded numerically as mild (1), moderate (2) to severe (3).
Time Frame: baseline, 4 months
Population: Participants completing the 4-month follow-up
Measure: Number; unit: participants
Arm/Group | Lidocaine | Botulinum
Number analyzed (Participants) | 7 | 9
participants | 3 | 4

4. Secondary Outcome: Clinical Response as Assessed by >20% Change From Baseline in Jaw Opening
Description: maximum mandibular range of motion scores (measured as the maximum interincisal distance and compensating for occlusion)
Time Frame: baseline, 4 months
Population: Participants completing the 4-month follow-up
Measure: Number; unit: participants
Arm/Group | Lidocaine | Botulinum
Number analyzed (Participants) | 7 | 9
participants | 2 | 0

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Lidocaine | Botulinum
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/10
Other Adverse Events (participants affected / at risk) | 1/7 | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine (N=7) | Botulinum (N=10)
Headache (General disorders) | 1 (1) | 1 (1)
facial muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes